CLINICAL TRIAL: NCT05571631
Title: Investigation of the Effect of the Combination of Arm Ergometer Exercise and Balance Training on Upper Extremity Function in People With Multiple Sclerosis
Brief Title: Effect of Arm Ergometer Exercise Training on Upper Extremity Function in People With Multiple Sclerosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Serkan Ozakbas, Prof. Dr., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7181-GOA
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; upper extremity; balance; rehabilitation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm ergometer-balance training (Experimental): Combination of arm ergometer exercise and balance training
  Interventions: Other: exercise
- arm ergometer (Experimental): Only arm ergometer exercise training
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Arm ergometer will aplied as an aerobic exercise. Combination of balance training and arm ergometer exerise program will applied.

SUMMARY:
This study will investigate the effects of a 12-week arm ergometer exercise and balance training on upper extremity function in persons with multiple sclerosis.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an inflammatory, demyelinating, neurodegenerative disease of the central nervous system of unknown etiology. The most common clinical signs and symptoms are motor dysfunction, fatigue, spasticity, impaired mobility, cognitive impairment, chronic pain, depression, decreased quality of life, and bladder and bowel dysfunction. 66% of people with MS (pwMS) have impaired upper extremity function.

As a result of the deterioration in upper extremity function, the performance of many daily living activities affects performance. As a result of this influence, there is a decrease in the functional independence of pwMS, quality of life and participation in activities in the community.

Another common symptom that reduces quality of life, independence, and participation in pwMS is balance disorder, seen in 75% of cases. Abnormality in balance control occurs due to lack of postural stability, limitation of stability limits, slowness to return to the starting position during bending and reaching activities. During interaction with the environment in daily life, proprioceptive inputs from the extremities and subsequent proper trunk control enable the person to keep the center of gravity on the support surface at rest and in activity. In this way, proximal stability is provided and tasks that require participation in daily life with distal mobility are performed. It is necessary to manage these progressive symptoms associated with the disease in order to increase the quality of life of pwMS, increase the rate of participation in society and maintain this increase.

Exercise training represents an existing behavioral treatment approach to safely manage many functional, symptomatic and quality-of-life outcomes in MS. Current literature reports that aerobic exercise has a positive effect on important parameters such as balance, fatigue, walking, quality of life, and pain in pwMS. At the same time, aerobic exercise training with arm ergometry allows pwMS to improve their upper extremity function. Apart from these, the literature has separately examined the effects of exercise training on upper extremity function and balance in pwMS, and positive effects have been shared separately. However, the relationship between these two important issues and the effect of exercise training on this relationship have not been examined.

The aim of the study is to examine the effects of exercise training on upper extremity function and balance in pwMS.

Persons who followed by the outpatient Multiple Sclerosis Clinic of Dokuz Eylül University Hospital will participate in the study. A total of 30 participants will randomly be divided into 2 groups as arm ergometer-balance training group and arm ergometer training group. Both exercise training will be given by a physiotherapist, supervised 2 days a week for 12 weeks. Assessments will done at baseline and after 12weeks (post-treatment). Assessments will be done by assessors who are blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

* A relapsing-remitting or secondary progressive type of multiple sclerosis,
* To be willing to participate in the study.

Exclusion Criteria:

* Another neurological disorder,
* Orthopedic surgery history including the elbow, wrist, shoulder, ankle-foot, knee, hip or spine, affecting balance and upper extremity functions,
* Diagnosed severe cognitive and/or psychiatric impairment,
* Having congestive heart failure, coronary, cerebrovascular, and pulmonary disease such as COPD
* Having cardiac disease such as hypertension that would be a contraindication to exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Nine-Hole Peg Test | Change from Baseline at 12 weeks
  The Nine-Hole Peg Test measures finger dexterity.

SECONDARY OUTCOMES:
Expanded Disability Status Scale | Baseline
  Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis. The Expanded Disability Status Scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Jamar Hand Dynamometer | Change from Baseline at 12 weeks
  The Jamar Hand Dynamometer will be used to measure isometric force and peak strength.
Arm Function in Multiple Sclerosis Questionnaire | Change from Baseline at 12 weeks
  Arm Function in Multiple Sclerosis Questionnaire is a unidimensional 31-item questionnaire for measuring arm function in MS. The total sum score ranged from 31 to 186 and a high score indicates a low degree of arm function.
Preference-based Multiple Sclerosis Index | Change from Baseline at 12 weeks
  The Preference-based Multiple Sclerosis Index is a brief patient-reported outcome measure of health-related quality of life that consists of 5 items: walking, fatigue, mood, concentration, and roles and responsibilities. The scoring algorithm ranges from 0 (dead) to 1 (perfect health).
Estimated VO2 Max | Change from Baseline at 12 weeks
  Estimated VO2max will be calculated Astrand-Rhyming Cycle Ergometer Test.
Modified Fatigue Impact Scale | Change from Baseline at 12 weeks
  The Modified Fatigue Impact Scale provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The scale consists of 21 items with Likert-type choose options. The total score for the scale is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items. The total score ranges from 0 to 84. A higher score indicates higher level of fatigue.
Timed Up and Go test | Change from Baseline at 12 weeks
  The Timed Up and Go test is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. During the test, the person is expected to wear their regular footwear and use any mobility aids that they would normally require. The time is calculated from the initiation of the instruction to start and ends when the patient has sit down. Higher time represents more static and dynamic balance and mobility impairment.
Activities-Specific Balance Confidence Scale | Change from Baseline at 12 weeks
  The Activities-Specific Balance Confidence Scale is a subjective measure of confidence in performing various ambulatory activities without falling or experiencing a sense of unsteadiness. 16-item self-report measure in which patients rate their balance confidence for performing activities. This stem is used to lead into each activity considered: "How confident are you that you will not lose your balance or become unsteady when you..." Items are rated on a rating scale that ranges from 0 - 100. Score of zero represents no confidence, a score of 100 represents complete confidence. Overall score is calculated by adding item scores and then dividing by the total number of items.
Coin Rotation Test | Change from Baseline at 12 weeks
  The coin Rotation Test is developed to assess fine motor skills and speed.

IPD SHARING:
Plan to Share IPD: Undecided